CLINICAL TRIAL: NCT02804243
Title: The Efficacy of Nasal High Flow Oxygen Therapy With Rehabilitation in the Patients With Chronic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hospital Organization Minami Kyoto Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 27-10
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2017-09

CONDITIONS: Chronic Respiratory Failure; Nasal High Flow Therapy; Rehabilitation; Exercise Endurance
Keywords: nasal high flow therapy; rehabilitation; exercise endurance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nasal high flow therapy (Active Comparator): In this group, patients have undergone rehabilitation under the nasal high flow therapy (FiO2 100%, oxygen flow from 30 to 60 L/min) during four weeks.
  Interventions: Device: nasal high flow therapy
- oxygen therapy (No Intervention): In this group, patients have undergone rehabilitation under the oxygen therapy via a nasal canula (6 L/min) during four weeks.

INTERVENTIONS:
Device: nasal high flow therapy — The nasal high flow therapy has enabled high flow oxygen to be derived through nasal cannula. This mode not only allows constant FiO2 during peak inspiratory flow but also confers benefits including a low level of continuous positive airway pressure with increased end-expiratory lung volume and reduced work of breathing, partly through intrinsic positive end-expiration pressure compensation and dead space washout. The inspired gases are warmed and humidified, improving comfort and possibly reducing airway inflammation, leading to improved drainage of respiratory secretions.
  Arms: nasal high flow therapy

SUMMARY:
The purpose of this study is to compare the exercise endurance between oxygen therapy with rehabilitation and nasal high flow therapy with rehabilitation for the patients with chronic respiratory failure receiving long-term oxygen therapy.

DETAILED DESCRIPTION:
In patients with chronic respiratory failure, pulmonary rehabilitation is recognized as an evidence-based treatment in improving exercise capacity, muscle strength, dyspnea, and quality of life. Oxygen supplementation during exercise induced dose-dependent improvement in endurance and symptom perception in chronic obstructive pulmonary disease patients. Recently, nasal high flow therapy which consists of high flow gas with an FiO2 ranging from 0.21 to nearly 1.0 adjusted by an oxygen blender, brought to body temperature, and saturated with water through an in-line humidifier is available.

The present study is randomised to compare the effect of exercise endurance between oxygen therapy with rehabilitation and nasal high flow therapy with rehabilitation for the patients with chronic respiratory failure receiving long-term oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic respiratory failure receiving long-term oxygen therapy for more than 3 months.

Exclusion Criteria:

* Subjects with severe cardiovascular disease, diabetes, neurological disease, and renal failure.
* Subject who are unable to undergo rehabilitation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Walk distance (measured by six minutes walking test) | Four weeks

SECONDARY OUTCOMES:
Six minutes walking test (minimum Oxygen Saturation of Arterial Blood Measured by Pulse Oximeter (SpO2) et.) | Four weeks
Exercise tolerance test (exercise time et.) | Four weeks
Body composition measured by InBody (muscle mass et.) | Four weeks
Arterial blood gas | Four weeks
Inflammation (CRP et.) | Four weeks
Nutritional status (body mass index(kg/m2) et.) | Four weeks
Sympathetic activity (Catecholamine et.) | Four weeks
Dyspnea (Modified Borg scale) | Four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Minami Kyoto Hospital, Jōyō, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chihara Y, Tsuboi T, Sumi K, Sato A. Effectiveness of high-flow nasal cannula on pulmonary rehabilitation in subjects with chronic respiratory failure. Respir Investig. 2022 Sep;60(5):658-666. doi: 10.1016/j.resinv.2022.05.002. Epub 2022 May 26. PMID 35644803